CLINICAL TRIAL: NCT03037034
Title: Novel Endoscopic Resection of Upper Gastrointestinal Subepithelial Tumors Originating From the Muscularis Propria: a Promising Forcep Strip Method
Brief Title: Novel Endoscopic Resection of Upper Gastrointestinal Subepithelial Tumors Originating From the Muscularis Propria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, In-Kyung Yoo, Clinical Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Novel Forcep Srip Method
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Subepithelial Tumor
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forcep Strip Method Treatment (Experimental): patients who have Gastrointestinal Subepithelial Tumors Originating from the Muscularis Propria are enrolled
  Interventions: Device: Forcep

INTERVENTIONS:
Device: Forcep — Following the injection around a submucosal tumor, the adjacent mucosa or submucosa was grasped with the forceps and pulled away to form a "tent". The tissue was dissected using an electrocoagulating current.

SUMMARY:
Endoscopic submucosal tumor resection using biopsy forceps was performed for 11 consecutive patients who had clinical indications for lesion removal. Following the injection around a submucosal tumor, the adjacent mucosa or submucosa was grasped with the forceps and pulled away to form a "tent". The tissue was dissected using an electrocoagulating current. In brief, the tumor was dissected from the muscularis propria layer and then carefully removed using forceps. Demographic data, indication for intervention, safety of the procedure and follow-up will be assessed.

DETAILED DESCRIPTION:
After the target lesion was identified, several marking dots were made around the lesion, using the hot biopsy forcep. A 0.9% saline solution mixed with epinephrine (1:10,000) and indigo carmine dye was injected along the border of the tumor to raise the gastric mucosa. Then, a circumferential incision was made along the margin of the targeted lesion, using the hot biopsy forceps, and the superficial mucosa was removed. Repeated injection was performed into the submucosal layer. The surrounding tissue was then carefully dissected using the hot biopsy forceps to the level of the deepest submucosal layer. The adjacent tissue was grasped using the forceps and pulled away, forming a "tent". To ensure complete resection, the muscular fibers and stalks that connected the tumor to the propria layer were shelled along the capsule of the tumor, using the coagulating forceps. The investigators used a coagulating forceps when strip the tissue of the outer longitudinal layer. Visible blood vessels in the submucosal layer were directly coagulated using coagulating forceps. After the lesion was removed, further visible blood vessels were coagulated. The hot biopsy forcep was used to apply a forced coagulation current (80 W, Effect 2, VIO300D; Erbe, Germany). However, coagulating forceps with a soft coagulation current (60 W, Effect 6, VIO300D; Erbe, Germany) were used to cut muscle fibers adjacent to the tumor or hemostasis.

ELIGIBILITY:
Inclusion Criteria:

1. the tumor size had increased on the follow up gastroscopy,
2. the EUS showed a well demarcated GI SET, or
3. they requested an endoscopic excision because the tumor was causing them anxiety.

Exclusion Criteria:

1. they had predominantly extraluminal growth,
2. they were ill demarcated, or
3. the EUS showed adjacent lymph nodes with a malignant appearance.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | 1 week
  Proportion of study patients with a histologically confirmed diagnosis after Forcep Strip Method

SECONDARY OUTCOMES:
The mean procedure time | 1day
  procedure time of submucosal tumor removal using forcep strip method
mean tumor size | 1day
  tumor size of submucosal tumor removed by forcep strip method
the mean hospitalization time | 1week
  patient hospitalization time during submucosal tumor removal
Adverse Events | 5 days
  Peri-interventional adverse events whether related or not
Tumor status after endoscopic resection | 10 months
  Local result during follow up after Forcep Strip Method

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Jai Chun, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Anamdong , Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No